CLINICAL TRIAL: NCT00715104
Title: An Open Label, Phase 2 Trial of Immunotherapy With Sipuleucel-T (Provenge®) as Neoadjuvant Treatment in Men With Localized Prostate Cancer
Brief Title: Sipuleucel-T as Neoadjuvant Treatment in Prostate Cancer
Acronym: NeoACT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dendreon (Industry)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P07-1
Record Dates: First submitted 2008-07-11; First posted 2008-07-15 (Estimated); Results first posted 2015-04-01 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — sipuleucel-T; Immunization, Secondary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sipuleucel-T with Booster (Experimental): Subjects were to receive 3 infusions of sipuleucel-T 12 weeks prior to RP, and then an additional booster infusion 13 weeks following RP.
  Interventions: Biological: Sipuleucel-T with Booster
- Sipuleucel-T without Booster (Experimental): Subjects were to receive 3 infusions of sipuleucel-T 12 weeks prior to RP, with no further sipuleucel-T treatment.
  Interventions: Biological: Sipuleucel-T without Booster

INTERVENTIONS:
Biological: Sipuleucel-T with Booster — Sipuleucel-T is an autologous active cellular immunotherapy product designed to stimulate an immune response against prostate cancer. Sipuleucel-T consists of autologous peripheral blood mononuclear cells (PBMCs), including antigen presenting cells (APCs), that have been activated in vitro with a recombinant fusion protein.
  Arms: Sipuleucel-T with Booster
Biological: Sipuleucel-T without Booster — Sipuleucel-T is an autologous active cellular immunotherapy product designed to stimulate an immune response against prostate cancer. Sipuleucel-T consists of autologous peripheral blood mononuclear cells (PBMCs), including antigen presenting cells (APCs), that have been activated in vitro with a recombinant fusion protein.
  Arms: Sipuleucel-T without Booster

SUMMARY:
This is an open label, Phase 2 trial of immunotherapy with sipuleucel-T as neoadjuvant treatment in men with localized prostate cancer.

DETAILED DESCRIPTION:
This is a single center, open label, Phase 2 study. Subjects will be treated with 3 infusions of sipuleucel-T prior to a scheduled radical prostatectomy (RP) surgery. To assess the immune response following treatment with sipuleucel-T, tissue from the prostatectomy specimen will be compared with tissue from the core biopsy specimen obtained prior to treatment with sipuleucel T. Following RP, subjects will be randomized to receive either a booster infusion of sipuleucel T or no further treatment with sipuleucel-T (i.e., booster: no booster).

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the prostate.
* Subject is scheduled for RP as the initial therapy for localized prostate cancer.
* Subject is ≥ 18 years of age.
* Subject has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Subject has adequate hematologic, renal, and liver function.

Exclusion Criteria:

* Subject has any evidence of metastasis.
* Subject received hormones, including luteinizing hormone-releasing hormone agonists, antiandrogens, or 5 α-reductase inhibitors at any time prior to study screening.
* Subject has received prior radiation therapy or chemotherapy for prostate cancer.
* Subject has received systemic steroid therapy within 14 days.
* Subject has a history of stage III or greater cancer, excluding prostate cancer.
* Subjects with a history of basal or squamous cell skin cancers are allowed, provided that the subject was adequately treated and is disease-free at the time of study screening.
* Subjects with a history of stage I or II cancer must have been adequately treated and been disease-free for ≥ 3 years prior to study screening.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-07; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andy Sandler, MD, Study Director — Dendreon
Locations (7):
- United States (7):
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Kaiser Permanente Portland, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - University of Utah School of Medicine, Salt Lake City, Utah
  - Virginia Mason Medical Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington

REFERENCES:
- [Derived] Sheikh N, Cham J, Zhang L, DeVries T, Letarte S, Pufnock J, Hamm D, Trager J, Fong L. Clonotypic Diversification of Intratumoral T Cells Following Sipuleucel-T Treatment in Prostate Cancer Subjects. Cancer Res. 2016 Jul 1;76(13):3711-8. doi: 10.1158/0008-5472.CAN-15-3173. Epub 2016 May 23. PMID 27216195
- See also: National Prostate Cancer Coalition — http://www.pcacoalition.org
- See also: USTOO International — http://www.ustoo.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted across 6 sites in the US. Screening and enrollment occurred from Sept 2008 - Dec 2012. 42 subjects were registered. 41 subjects received at least 1 sipuleucel-T infusion prior to radical prostatectomr (RP),18 subjects were randomized to the booster group,15 were randomized to the no booster group; and 8 were not randomized.
Groups:
- Sipuleucel-T Without Randomization to Booster: Subjects were to receive 3 infusions of sipuleucel-T 12 weeks prior to RP, and declined participation in the post-RP booster phase (received no further sipuleucel-T treatment).
Period: Overall Study
Arm/Group | Sipuleucel-T With Booster | Sipuleucel-T Without Booster | Sipuleucel-T Without Randomization to Booster
Started | 18 | 16 | 8
Completed | 18 | 16 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sipuleucel-T With Booster: Subjects received 3 infusions of sipuleucel-T 12 weeks prior to RP, and then an additional booster infusion 13 weeks following RP.
- Sipuleucel-T Without Booster: Subjects received 3 infusions of sipuleucel-T 12 weeks prior to RP, with no further sipuleucel-T treatment.
- Sipuleucel-T Without Randomization to Booster: Subjects received 3 infusions of sipuleucel-T 12 weeks prior to RP, and declined participation in the post-RP booster phase(received no further sipuleucel-T treatment).
- Total: Total of all reporting groups
Arm/Group | Sipuleucel-T With Booster | Sipuleucel-T Without Booster | Sipuleucel-T Without Randomization to Booster | Total
Number analyzed (Participants) | 18 | 16 | 8 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 12 | 5 | 31
  >=65 years | 4 | 4 | 3 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (5.6) | 61.4 (5.3) | 62.1 (5.7) | 61.1 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 18 | 16 | 8 | 42
Region of Enrollment [Number; unit: participants]
  United States | 18 | 16 | 8 | 42

OUTCOME MEASURES:

1. Primary Outcome: Change in the Number of Infiltrating CD3+ T Cells Within the Prostate Tissue Between the Biopsy and the Post-RP Tissue Specimens in Each Subject
Description: CD3+ T cell infiltration within prostate tissue was quantified using immunohistochemistry (IHC) staining techniques. Cells were enumerated per unit area (cells/μm2). For post-RP tissue specimens, three areas of interest were identified: Benign tissue, tumor tissue, and tumor interface tissue.
Time Frame: Pre-treatment biopsy (baseline) and post-RP (12 weeks post-treatment)
Population: All subjects who received at least 1 infusion of sipuleucel-T and underwent subsequent RP.
  Results are not presented by arm because all assessments were performed prior to randomization to booster.
Measure: Mean (Standard Error); unit: cells/μm2
Groups:
- Biopsy Benign Tissue: Tissue from the core biopsy specimen obtained prior to treatment with sipuleucel-T
- Post-RP Benign Tissue: Benign tissue from post-treatment with sipuleucel-T and post-RP
- Post-RP Tumor Tissue: Tumor tissue from post-treatment with sipuleucel-T and post-RP
- Post-RP Tumor Interface: Tumor interface (the junction of normal and malignant) tissue from post-treatment with sipuleucel-T and post-RP
Arm/Group | Biopsy Benign Tissue | Post-RP Benign Tissue | Post-RP Tumor Tissue | Post-RP Tumor Interface
Number analyzed (Participants) | 37 | 37 | 37 | 37
cells/μm2 | 2.33 (0.34) | 2.03 (0.19) | 1.98 (0.18) | 6.39 (0.61)
Statistical Analysis 1: Comparison: Biopsy Benign Tissue vs Post-RP Benign Tissue; A 2-fold increase in CD3+ T cell counts from biopsy to post-RP was considered a positive response. The number of infiltrating CD3+ T cells/μm2 was coded as binary with each subject categorized as having at least a 2-fold increase from baseline or not. One sample Chi-square test for a binary response, with a null hypothesis of 15% was implemented. The tests were done using post-treatment post-RP benign tissue, tumor tissue, and tumor interface compared to the biopsy benign tissue; Test type: Superiority or Other; p = 1.000, Chi-squared — Bonferroni-adjusted p-values will be reported to alleviate the multiple testing problem; pbon = minimum of p*3 and 1 (p = the nominal p-value from the test, pbon = the Bonferroni-adjusted p-value). Confidence intervals will be adjusted similarly; % Subjects with 2-fold increase = 16.2, 95% CI 2-sided [1.7 to 30.7]
Statistical Analysis 2: Comparison: Biopsy Benign Tissue vs Post-RP Tumor Tissue; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 1.000, Chi-squared — [p-value comment as in outcome 1, analysis 1]; % Subjects with 2-fold increase = 18.9, 95% CI 2-sided [3.5 to 34.3]
Statistical Analysis 3: Comparison: Biopsy Benign Tissue vs Post-RP Tumor Interface; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Chi-squared — [p-value comment as in outcome 1, analysis 1]; % Subjects with 2-fold increase = 70.3, 95% CI 2-sided [52.3 to 88.3]

2. Secondary Outcome: Change in the Number of Infiltrating CD4+ T Cells Within the Prostate Tissue Between the Biopsy and the Post-RP Tissue Specimens in Each Subject
Description: CD4+ T cell infiltration within prostate tissue was quantified using immunohistochemistry (IHC) staining techniques. Cells were enumerated per unit area (cells/μm2). For post-RP tissue specimens, three areas of interest were identified: Benign tissue, tumor tissue, and tumor interface tissue.
Time Frame: Pre-treatment biopsy (baseline) and post-RP (12 weeks post-treatment)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: cells/μm2
Groups:
- Post-RP Tumor Interface Tissue: Tumor interface (the junction of normal and malignant) tissue from post-treatment with sipuleucel-T and post-RP
Arm/Group | Biopsy Benign Tissue | Post-RP Benign Tissue | Post-RP Tumor Tissue | Post-RP Tumor Interface Tissue
Number analyzed (Participants) | 36 | 36 | 36 | 36
cells/μm2 | 0.93 (0.24) | 0.43 (0.09) | 0.74 (0.13) | 3.83 (0.49)
Statistical Analysis 1: Comparison: Biopsy Benign Tissue vs Post-RP Benign Tissue; A 2-fold increase in CD4+ T cell counts from biopsy to post-RP was considered a positive response. The number of infiltrating CD4+ T cells/μm2 was coded as binary with each subject categorized as having at least a 2-fold increase from baseline or not. One sample Chi-square test for a binary response, with a null hypothesis of 15% was implemented. The tests were done using post-treatment post-RP benign tissue, tumor tissue, and tumor interface compared to the biopsy benign tissue; Test type: Superiority or Other; p = 1.000, Chi-squared — [p-value comment as in outcome 1, analysis 1]; % subjects with 2-fold increase = 20.6, 95% CI 2-sided [4.0 to 37.2]
Statistical Analysis 2: Comparison: Biopsy Benign Tissue vs Post-RP Tumor Tissue; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.014, Chi-squared — [p-value comment as in outcome 1, analysis 1]; % subjects with 2-fold increase = 32.4, 95% CI 2-sided [13.1 to 51.6]
Statistical Analysis 3: Comparison: Biopsy Benign Tissue vs Post-RP Tumor Interface Tissue; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Chi-squared — [p-value comment as in outcome 1, analysis 1]; % subjects with 2-fold increase = 79.4, 95% CI 2-sided [62.8 to 96.0]

3. Secondary Outcome: Change in the Number of Infiltrating CD8+ T Cells Within the Prostate Tissue Between the Biopsy and the Post-RP Tissue Specimens in Each Subject
Description: CD8+ T cell infiltration within prostate tissue was quantified using immunohistochemistry (IHC) staining techniques. Cells were enumerated per unit area (cells/μm2). For post-RP tissue specimens, three areas of interest were identified: Benign tissue, tumor tissue, and tumor interface tissue.
Time Frame: Pre-treatment biopsy (baseline) and post-RP (12 weeks following sipuleucel-T)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: cells/μm2
Arm/Group | Biopsy Benign Tissue | Post-RP Benign Tissue | Post-RP Tumor Tissue | Post-RP Tumor Interface Tissue
Number analyzed (Participants) | 37 | 37 | 37 | 37
cells/μm2 | 0.65 (0.08) | 0.94 (0.14) | 0.88 (0.12) | 2.87 (0.25)
Statistical Analysis 1: Comparison: Biopsy Benign Tissue vs Post-RP Benign Tissue; A 2-fold increase in CD8+ T cell counts from biopsy to post-RP was considered a positive response. The number of infiltrating CD8+ T cells/μm2 was coded as binary with each subject categorized as having at least a 2-fold increase from baseline or not. One sample Chi-square test for a binary response, with a null hypothesis of 15% was implemented. The tests were done using post-treatment post-RP benign tissue, tumor tissue, and tumor interface compared to the biopsy benign tissue; Test type: Superiority or Other; p = 0.002, Chi-squared — [p-value comment as in outcome 1, analysis 1]; % subjects with 2-fold increase = 35.1, 95% CI 2-sided [16.3 to 53.9]
Statistical Analysis 2: Comparison: Biopsy Benign Tissue vs Post-RP Tumor Tissue; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.036, Chi-squared — [p-value comment as in outcome 1, analysis 1]; % subjects with 2-fold increase = 29.7, 95% CI 2-sided [11.7 to 47.7]
Statistical Analysis 3: Comparison: Biopsy Benign Tissue vs Post-RP Tumor Interface Tissue; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Chi-squared — [p-value comment as in outcome 1, analysis 1]; % subjects with 2-fold increase = 83.8, 95% CI 2-sided [69.3 to 98.3]

4. Secondary Outcome: Change in Antigen PA2024-specific T Cell Immunity in Peripheral Blood
Description: Antigen PA2024-specific T cell immune response is measured using interferon gamma (IFN-γ) enzyme-linked immunospot (ELISPOT) assays.
  This analysis was performed as previously described in Fong L et al. (J Immunol. 2001;167(12):7150-7156.). The unit of analysis is the number of IFN-γ ELISPOT counts per 300,000 peripheral blood mononuclear cells.
Time Frame: Baseline (screening visit) and up to 12-weeks post-RP visit (24 weeks following sipuleucel-T)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: numbers of spots
Groups:
- Baseline: ELISPOT for PA2024 at baseline
- Pre-RP Visit: ELISPOT for PA2024 at Pre-RP Visit
- 6 Weeks Post-RP: ELISPOT for PA2024 at 6 Weeks post-RP
- 12 Weeks Post-RP: ELISPOT for PA2024 at 12 Weeks post-RP
Arm/Group | Baseline | Pre-RP Visit | 6 Weeks Post-RP | 12 Weeks Post-RP
Number analyzed (Participants) | 33 | 28 | 23 | 29
numbers of spots | 4.9 (2.4) | 56.6 (14.9) | 26.5 (9.1) | 52.3 (17.6)
Statistical Analysis 1: Comparison: Baseline vs Pre-RP Visit vs 6 Weeks Post-RP vs 12 Weeks Post-RP; The change over time was evaluated by using repeated measure analysis of variance (ANOVA) methods with a mixed model approach. The ranked data were used in the statistical model; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P value is for the visit effect in the mixed model; Randomization groups, visits (up to 12-weeks Post-RP), and randomization groups × visits interaction were included in the mixed model

5. Secondary Outcome: Change in Antigen PAP-specific T Cell Immunity in Peripheral Blood
Description: Antigen PAP-specific T cell immune response is measured using interferon gamma (IFN-γ) enzyme-linked immunospot (ELISPOT) assays. PAP = Prostatic Acid Phosphatase.
Time Frame: Baseline (screening visit) and up to 12-weeks post-RP visit (24 months post sipuleucel-T)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: numbers of spots
Groups:
- Baseline: ELISPOT for PAP at baseline
- Pre-RP Visit: ELISPOT for PAP at pre-RP visit
- 6 Weeks Post-RP: ELISPOT for PAP at 6 Weeks post-RP
- 12 Weeks Post-RP: ELISPOT for PAP at 12 Weeks post-RP
Arm/Group | Baseline | Pre-RP Visit | 6 Weeks Post-RP | 12 Weeks Post-RP
Number analyzed (Participants) | 33 | 28 | 23 | 29
numbers of spots | 2.2 (1.7) | 13.3 (4.9) | 2.0 (1.2) | 12.8 (5.6)
Statistical Analysis 1: Comparison: Baseline vs Pre-RP Visit vs 6 Weeks Post-RP vs 12 Weeks Post-RP; Repeated measure analysis of variance (ANOVA) methods with a mixed model approach was used. The ranked data were used in the statistical model; Test type: Superiority or Other; p = 0.173, Mixed Models Analysis — P value is for the visit effect in the mixed model; [statistical method as in outcome 4, analysis 1]

6. Secondary Outcome: Effect of a Post-RP Booster Infusion of Sipuleucel-T Over Time of Antigen PA2024-Specific T Cell Immunity in the Peripheral Blood.
Description: The number of PA2024-specific T cells was enumerated by interferon gamma (IFN-γ) enzyme-linked immunospot (ELISPOT) assays (memory T cells).
Time Frame: 12 Weeks Post-RP (Pre-booster) and up to 72 Weeks post-RP
Population: Subjects received at least 1 infusion of sipuleucel-T, were randomized to receive a booster, and had blood samples suitable for ELISPOT analysis.
Measure: Mean (Standard Error); unit: numbers of spots
Groups:
- 12 Weeks Post-RP/Pre-Booster: ELISPOT for PA2024 measured at 12 Weeks Post-RP/Pre-Booster for subjects randomized to booster
- 24 Weeks Post-RP: ELISPOT for PA2024 measured at 24 Weeks Post-RP for subjects randomized to booster
- 48 Weeks Post-RP: ELISPOT for PA2024 measured at 48 Weeks Post-RP for subjects randomized to booster
- 72 Weeks Post-RP: ELISPOT for PA2024 measured at 72 Weeks Post-RP for subjects randomized to booster
Arm/Group | 12 Weeks Post-RP/Pre-Booster | 24 Weeks Post-RP | 48 Weeks Post-RP | 72 Weeks Post-RP
Number analyzed (Participants) | 16 | 12 | 13 | 10
numbers of spots | 35.6 (14.9) | 25.6 (9.7) | 23.5 (13.1) | 18.0 (5.0)
Statistical Analysis 1: Comparison: 12 Weeks Post-RP/Pre-Booster vs 24 Weeks Post-RP; The change over time was evaluated by using repeated measure analysis of variance (ANOVA) methods with a mixed model approach to allow for a varying number of follow-up measurements. The ranked data were used in the statistical model; Test type: Superiority or Other; p = 0.667, Mixed Models Analysis — P value compares 24 week post-RP to pre-booster (12 weeks post RP)
Statistical Analysis 2: Comparison: 12 Weeks Post-RP/Pre-Booster vs 48 Weeks Post-RP; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.191, Mixed Models Analysis — P value compares 48 week post-RP to pre-booster (12 weeks post RP)
Statistical Analysis 3: Comparison: 12 Weeks Post-RP/Pre-Booster vs 72 Weeks Post-RP; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.699, Mixed Models Analysis — P value compares 72 week post-RP to pre-booster (12 weeks post RP)

7. Secondary Outcome: Effect of a Post-RP Booster Infusion of Sipuleucel-T Over Time of Antigen PAP-Specific T Cell Immunity in the Peripheral Blood.
Description: The number of PAP-specific T cells was enumerated by interferon gamma (IFN-γ) enzyme-linked immunospot (ELISPOT) assays (memory T cells). PAP = Prostatic Acid Phosphatase.
Time Frame: 12 Weeks Post-RP (Pre-booster) and up to 72 Weeks post-RP
Population: as for outcome 6
Measure: Mean (Standard Error); unit: number of spots
Groups:
- 12 Weeks Post-RP/Pre-Booster: ELISPOT for PAP measured at 12 Weeks Post-RP/Pre-Booster for subjects randomized to booster
- 24 Weeks Post-RP: ELISPOT for PAP measured at 24 Weeks Post-RP for subjects randomized to booster
- 48 Weeks Post-RP: ELISPOT for PAP measured at 48 Weeks Post-RP for subjects randomized to booster
- 72 Weeks Post-RP: ELISPOT for PAP measured at 72 Weeks Post-RP for subjects randomized to booster
Arm/Group | 12 Weeks Post-RP/Pre-Booster | 24 Weeks Post-RP | 48 Weeks Post-RP | 72 Weeks Post-RP
Number analyzed (Participants) | 16 | 12 | 13 | 10
number of spots | 9.2 (5.4) | 0.3 (0.9) | 6.2 (4.8) | 0.4 (1.0)
Statistical Analysis 1: Comparison: 12 Weeks Post-RP/Pre-Booster vs 24 Weeks Post-RP; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.086, Mixed Models Analysis — P value compares 24 week post-RP to pre-booster (12 weeks post RP)
Statistical Analysis 2: Comparison: 12 Weeks Post-RP/Pre-Booster vs 48 Weeks Post-RP; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.432, Mixed Models Analysis — P value compares 48 week post-RP to pre-booster (12 weeks post RP)
Statistical Analysis 3: Comparison: 12 Weeks Post-RP/Pre-Booster vs 72 Weeks Post-RP; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.249, Mixed Models Analysis — P value compares 72 week post-RP to pre-booster (12 weeks post RP)

8. Secondary Outcome: Comparison of Booster Effect in Antigen PA2024-Specific T Cell Immunity Over Time Between the Two Randomized Groups
Description: The number of Antigen PA2024-specific T cells was enumerated by interferon gamma (IFN-γ) enzyme-linked immunospot (ELISPOT) assays (memory T cells). The two groups were compared in the statistical model are: Randomized to Booster and Randomized to No Booster.
Time Frame: 12 Weeks Post-RP (Pre-booster) and up to 72 Weeks post-RP
Population: Subjects received at least 1 infusion of sipuleucel-T, were randomized to receive either a booster infusion or no further treatment following RP, and had blood samples suitable for ELISPOT analysis.
Measure: Mean (Standard Error); unit: number of spots
Groups:
- Booster: 12 Weeks Post-RP/Pre-Booster: ELISPOT for PA2024 measured at 12 Weeks Post-RP/Pre-Booster for subjects randomized to booster
- No Booster: 12 Weeks Post-RP/Pre-Booster: ELISPOT for PA2024 measured at 12 Weeks Post-RP/Pre-Booster for subjects randomized to no booster
- Booster: 24 Weeks Post-RP: ELISPOT for PA2024 measured at 24 Weeks Post-RP for subjects randomized to booster
- No Booster: 24 Weeks Post-RP: ELISPOT for PA2024 measured at 24 Weeks Post-RP for subjects randomized to no booster
- Booster: 48 Weeks Post-RP: ELISPOT for PA2024 measured at 48 Weeks Post-RP for subjects randomized to booster
- No Booster: 48 Weeks Post-RP: ELISPOT for PA2024 measured at 48 Weeks Post-RP for subjects randomized to no booster
- Booster: 72 Weeks Post-RP: ELISPOT for PA2024 measured at 72 Weeks Post-RP for subjects randomized to booster
- No Booster: 72 Weeks Post-RP: ELISPOT for PA2024 measured at 72 Weeks Post-RP for subjects randomized to no booster
Arm/Group | Booster: 12 Weeks Post-RP/Pre-Booster | No Booster: 12 Weeks Post-RP/Pre-Booster | Booster: 24 Weeks Post-RP | No Booster: 24 Weeks Post-RP | Booster: 48 Weeks Post-RP | No Booster: 48 Weeks Post-RP | Booster: 72 Weeks Post-RP | No Booster: 72 Weeks Post-RP
Number analyzed (Participants) | 16 | 10 | 12 | 12 | 13 | 11 | 10 | 14
number of spots | 35.6 (14.9) | 81.7 (44.4) | 25.6 (9.7) | 22.3 (9.2) | 23.5 (13.1) | 19.5 (9.3) | 18.0 (5.0) | 12.6 (3.7)
Statistical Analysis 1: Comparison: Booster: 12 Weeks Post-RP/Pre-Booster vs No Booster: 12 Weeks Post-RP/Pre-Booster vs Booster: 24 Weeks Post-RP vs No Booster: 24 Weeks Post-RP vs Booster: 48 Weeks Post-RP vs No Booster: 48 Weeks Post-RP vs Booster: 72 Weeks Post-RP vs No Booster: 72 Weeks Post-RP; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.950, Mixed Models Analysis — P value is based on the treatment effect in the mixed model; Mixed model includes randomization group, visit, and randomization group × visit interaction, with subject as a random effect

9. Secondary Outcome: Comparison of Booster Effect in Antigen PAP-Specific T Cell Immunity Over Time Between the Two Randomized Groups
Description: The number of Antigen PAP-specific T cells was enumerated by interferon gamma (IFN-γ) enzyme-linked immunospot (ELISPOT) assays (memory T cells). The two groups were compared in the statistical model are: Randomized to Booster and Randomized to No Booster. PAP = Prostatic Acid Phosphatase.
Time Frame: 12 Weeks Post-RP (Pre-booster) and up to 72 Weeks post-RP
Population: as for outcome 8
Measure: Mean (Standard Error); unit: numbers of spots
Groups:
- Booster: 12 Weeks Post-RP/Pre-Booster: ELISPOT for PAP measured at 12 Weeks Post-RP/Pre-Booster for subjects randomized to booster
- No Booster: 12 Weeks Post-RP/Pre-Booster: ELISPOT for PAP measured at 12 Weeks Post-RP/Pre-Booster for subjects randomized to no booster
- Booster: 24 Weeks Post-RP: ELISPOT for PAP measured at 24 Weeks Post-RP for subjects randomized to booster
- No Booster: 24 Weeks Post-RP: ELISPOT for PAP measured at 24 Weeks Post-RP for subjects randomized to no booster
- Booster: 48 Weeks Post-RP: ELISPOT for PAP measured at 48 Weeks Post-RP for subjects randomized to booster
- No Booster: 48 Weeks Post-RP: ELISPOT for PAP measured at 48 Weeks Post-RP for subjects randomized to no booster
- Booster: 72 Weeks Post-RP: ELISPOT for PAP measured at 72 Weeks Post-RP for subjects randomized to booster
- No Booster: 72 Weeks Post-RP: ELISPOT for PAP measured at 72 Weeks Post-RP for subjects randomized to no booster
Arm/Group | Booster: 12 Weeks Post-RP/Pre-Booster | No Booster: 12 Weeks Post-RP/Pre-Booster | Booster: 24 Weeks Post-RP | No Booster: 24 Weeks Post-RP | Booster: 48 Weeks Post-RP | No Booster: 48 Weeks Post-RP | Booster: 72 Weeks Post-RP | No Booster: 72 Weeks Post-RP
Number analyzed (Participants) | 16 | 10 | 12 | 12 | 13 | 11 | 10 | 14
numbers of spots | 9.2 (5.4) | 20.2 (13.9) | 0.3 (0.9) | 4.8 (1.6) | 6.2 (4.8) | 2.7 (1.7) | 0.4 (1.0) | 1.9 (1.7)
Statistical Analysis 1: Comparison: Booster: 12 Weeks Post-RP/Pre-Booster vs No Booster: 12 Weeks Post-RP/Pre-Booster vs Booster: 24 Weeks Post-RP vs No Booster: 24 Weeks Post-RP vs Booster: 48 Weeks Post-RP vs No Booster: 48 Weeks Post-RP vs Booster: 72 Weeks Post-RP vs No Booster: 72 Weeks Post-RP; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.048, Mixed Models Analysis — P value is based on the treatment effect in the mixed model; [statistical method as in outcome 8, analysis 1]

ADVERSE EVENTS:
Groups:
- Sipuleucel-T With Booster: Subjects receive 3 infusions of sipuleucel-T 12 weeks prior to RP, and then received an additional booster infusion 13 weeks after RP.
- Sipuleucel-T Without Randomization to Booster: Subjects received 3 infusions of sipuleucel-T 12 weeks prior to RP, and declined participation in the post-RP booster phase (received no further sipuleucel-T treatment).
Arm/Group | Sipuleucel-T With Booster | Sipuleucel-T Without Booster | Sipuleucel-T Without Randomization to Booster
Serious Adverse Events (participants affected / at risk) | 1/18 | 4/16 | 1/8
Other Adverse Events (participants affected / at risk) | 18/18 | 14/16 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sipuleucel-T With Booster (N=18) | Sipuleucel-T Without Booster (N=16) | Sipuleucel-T Without Randomization to Booster (N=8)
ARRHYTHMIA (Cardiac disorders) | 0 | 1 | 0
RETINAL VEIN OCCLUSION (Eye disorders) | 1 | 0 | 0
VISION BLURRED (Eye disorders) | 0 | 1 | 0
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 0 | 1 | 0
B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
DIZZINESS (Nervous system disorders) | 0 | 1 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 1 | 0
DISORIENTATION (Psychiatric disorders) | 0 | 1 | 0
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sipuleucel-T With Booster (N=18) | Sipuleucel-T Without Booster (N=16) | Sipuleucel-T Without Randomization to Booster (N=8)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 | 1 | 0
CARDIAC FLUTTER (Cardiac disorders) | 0 | 1 | 0
PALPITATIONS (Cardiac disorders) | 0 | 0 | 1
CONJUNCTIVITIS (Eye disorders) | 1 | 1 | 0
EYE SWELLING (Eye disorders) | 0 | 1 | 0
SCLERAL HAEMORRHAGE (Eye disorders) | 0 | 1 | 0
VITREOUS DETACHMENT (Eye disorders) | 1 | 0 | 0
VITREOUS HAEMORRHAGE (Eye disorders) | 2 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 0 | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 2 | 2 | 2
DYSPEPSIA (Gastrointestinal disorders) | 2 | 0 | 0
FOOD POISONING (Gastrointestinal disorders) | 0 | 0 | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 4 | 2 | 1
UMBILICAL HERNIA (Gastrointestinal disorders) | 1 | 0 | 0
VOMITING (Gastrointestinal disorders) | 2 | 1 | 0
ASTHENIA (General disorders) | 2 | 0 | 0
AXILLARY PAIN (General disorders) | 0 | 0 | 1
CHEST PAIN (General disorders) | 0 | 0 | 1
CHILLS (General disorders) | 4 | 1 | 0
FATIGUE (General disorders) | 9 | 8 | 5
FEELING JITTERY (General disorders) | 0 | 1 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 1 | 1 | 1
INFUSION SITE ERYTHEMA (General disorders) | 0 | 0 | 1
INFUSION SITE IRRITATION (General disorders) | 0 | 1 | 0
INFUSION SITE PAIN (General disorders) | 0 | 0 | 1
INJECTION SITE EXTRAVASATION (General disorders) | 0 | 1 | 1
INJECTION SITE PRURITUS (General disorders) | 0 | 1 | 0
MALAISE (General disorders) | 1 | 1 | 1
OEDEMA PERIPHERAL (General disorders) | 0 | 1 | 0
PAIN (General disorders) | 0 | 1 | 0
PYREXIA (General disorders) | 2 | 0 | 0
THROMBOSIS IN DEVICE (General disorders) | 1 | 0 | 0
BRONCHITIS (Infections and infestations) | 0 | 1 | 0
CELLULITIS (Infections and infestations) | 0 | 0 | 1
INFECTION (Infections and infestations) | 0 | 1 | 0
INFLUENZA (Infections and infestations) | 1 | 1 | 0
NASOPHARYNGITIS (Infections and infestations) | 2 | 1 | 1
ORCHITIS (Infections and infestations) | 1 | 0 | 0
SINUSITIS (Infections and infestations) | 0 | 1 | 0
SKIN INFECTION (Infections and infestations) | 1 | 0 | 0
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 | 1 | 0
TOOTH INFECTION (Infections and infestations) | 2 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 | 3 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 2 | 1
CITRATE TOXICITY (Injury, poisoning and procedural complications) | 2 | 4 | 2
CONTUSION (Injury, poisoning and procedural complications) | 2 | 3 | 0
EYE INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 1 | 0
GASTROENTERITIS RADIATION (Injury, poisoning and procedural complications) | 1 | 0 | 0
JOINT INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0
PERIORBITAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 1 | 0
TOOTH INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 2 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 2 | 0
BLOOD PRESSURE DECREASED (Investigations) | 1 | 0 | 0
HAEMATOCRIT DECREASED (Investigations) | 1 | 0 | 0
HAEMOGLOBIN DECREASED (Investigations) | 1 | 0 | 0
WEIGHT INCREASED (Investigations) | 1 | 0 | 0
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 | 0 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 1 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 2 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 1 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 | 4 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
TENOSYNOVITIS STENOSANS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
HEPATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
MELANOCYTIC NAEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
DISTURBANCE IN ATTENTION (Nervous system disorders) | 1 | 0 | 0
DIZZINESS (Nervous system disorders) | 2 | 0 | 1
HEADACHE (Nervous system disorders) | 6 | 4 | 0
HYPOAESTHESIA (Nervous system disorders) | 1 | 0 | 0
MIGRAINE (Nervous system disorders) | 0 | 1 | 0
PARAESTHESIA (Nervous system disorders) | 1 | 0 | 2
PARAESTHESIA ORAL (Nervous system disorders) | 6 | 4 | 1
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 | 0 | 1
PRESYNCOPE (Nervous system disorders) | 2 | 0 | 0
RADICULITIS LUMBOSACRAL (Nervous system disorders) | 1 | 0 | 0
SYNCOPE (Nervous system disorders) | 0 | 1 | 0
TREMOR (Nervous system disorders) | 0 | 1 | 0
PERINEAL HAEMATOMA (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
ANXIETY (Psychiatric disorders) | 2 | 1 | 0
DEPRESSION (Psychiatric disorders) | 0 | 1 | 0
INSOMNIA (Psychiatric disorders) | 2 | 0 | 0
LIBIDO DECREASED (Psychiatric disorders) | 1 | 0 | 0
CALCULUS BLADDER (Renal and urinary disorders) | 0 | 1 | 0
DYSURIA (Renal and urinary disorders) | 0 | 1 | 1
NOCTURIA (Renal and urinary disorders) | 1 | 0 | 0
POLLAKIURIA (Renal and urinary disorders) | 1 | 0 | 0
URINARY INCONTINENCE (Renal and urinary disorders) | 0 | 1 | 0
URINE ODOUR ABNORMAL (Renal and urinary disorders) | 0 | 1 | 0
GYNAECOMASTIA (Reproductive system and breast disorders) | 0 | 1 | 0
HAEMATOSPERMIA (Reproductive system and breast disorders) | 0 | 0 | 1
PENILE PAIN (Reproductive system and breast disorders) | 0 | 0 | 1
PERINEAL PAIN (Reproductive system and breast disorders) | 1 | 0 | 0
TESTICULAR PAIN (Reproductive system and breast disorders) | 0 | 2 | 0
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
RESPIRATORY DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
SNORING (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
BLISTER (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
HAIR GROWTH ABNORMAL (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
FLUSHING (Vascular disorders) | 1 | 0 | 1
HOT FLUSH (Vascular disorders) | 2 | 3 | 0
HYPERTENSION (Vascular disorders) | 2 | 0 | 0
HYPOTENSION (Vascular disorders) | 1 | 0 | 0
PHLEBITIS (Vascular disorders) | 0 | 0 | 1
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study will be published and/or presented in an integrated manner reflecting the results observed across all participating centers. Accordingly, decisions on timing and content of publications and presentations relating to the study will be coordinated by Dendreon in communication with institutions contributing patients to the study.